CLINICAL TRIAL: NCT05038813
Title: A Single-arm, Multi-center Exploratory Clinical Study of Anlotinib Combined With TQB2450 (PD-L1 Inhibitor) in the Treatment of Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Anlotinib Combined With TQB2450 (PD-L1 Inhibitor) in the Treatment of Advanced Esophageal Squamous Cell Carcinoma(ESCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-E-003
Record Dates: First submitted 2021-09-06; First posted 2021-09-09 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib combined with TQB2450 (Experimental): Anlotinib: 12mg, capsule, once a day. TQB2450: 1200mg, Injection, Once every three weeks.
  Interventions: Drug: Anlotinib+TQB2450

INTERVENTIONS:
Drug: Anlotinib+TQB2450 — Anlotinib: 12mg, orally once a day (orally before breakfast, the daily medication time should be as the same as possible), continuous taking for 2 weeks, stopping for 1 week, 3 weeks (21 days) as a treatment cycle, until the disease progresses or Intolerable.
  TQB2450: 1200mg, diluted to 250mL with normal saline, infusion time 60±10mins. The medication is taken on the first day of each cycle, and 3 weeks (21 days) is a treatment cycle. Until the emergence of disease progression or intolerable toxicity, the longest use time does not exceed 24 months.

SUMMARY:
To evaluate the effectiveness and safety of anlotinib combined with TQB2450 (PD-L1 inhibitor) in the first-line treatment of patients with advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with the follow-up.
* Unresectable locally advanced, unresectable recurrent or metastatic ESCC confirmed by histopathology (excluding mixed adenosquamous carcinoma);
* Patients who have not received systemic treatment in the past, or who have previously received (neo) adjuvant treatment/radical treatment programs (including radical surgical resection and radical radiotherapy and chemotherapy programs) who have relapsed for more than 6 months; Note: Including patients with advanced or recurring non-target lesions who have progressed again after simple radiotherapy. For local lesions (non-target lesions), the time from the end of palliative treatment to the enrollment time is> 2 weeks;
* According to the RECIST version 1.1 of the curative effect evaluation standard for solid tumors, there is at least one measurable lesion, and it can be accurately measured by magnetic resonance imaging (MRI) or computed tomography (CT) in at least one direction (the largest diameter needs to be recorded) , Where the longest diameter at baseline is ≥10 mm (if it is a lymph node, the short diameter is required to be ≥15 mm); the measurable lesions should not have received local treatment such as radiotherapy (the lesions located in the previous radiotherapy area, if it is confirmed to have progressed, and meet RECIST1.1 standard, target lesions can also be selected);
* Male or female patients between 18-75 years old;
* Eastern Cooperative Oncology Group (ECOG) physical status (PS) score: 0-1 points;
* The estimated survival period exceeds 3 months;
* Possess sufficient organ and bone marrow function, that is, meet the following standards:

  1. Routine blood examination standards must be met (no blood transfusion and blood products within 14 days, no correction with G-CSF and other hematopoietic stimulating factors):Hemoglobin content (HB) ≥100g/L; White blood cell content (WBC) ≥3.0×10^9/L; Neutrophil count (ANC)≥1.5×10^9/L; Platelet count (PLT) ≥75×10^9/L.
  2. The biochemical inspection shall meet the following standards:Total serum bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); ALT and AST≤2.5ULN; if there is liver metastasis, ALT and AST≤5ULN;Cr≤1.5ULN or creatinine clearance rate (CCr)≥60ml/min, (Cockcroft-Gault formula).
  3. Adequate coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN;
  4. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%);
  5. Myocardial enzyme spectrum: within the normal range.
* Women of childbearing age must take appropriate contraceptive measures from screening to 3 months after stopping the study treatment, and participants must be non-lactating patients. Before starting the administration, the pregnancy test is negative, or meeting one of the following criteria proves that there is no risk of pregnancy:

  1. Postmenopausal is defined as amenorrhea at least 12 months after the age is over 50 years and all exogenous hormone replacement therapy is stopped;
  2. For women younger than 50 years old, if the amenorrhea is 12 months or more after stopping all exogenous hormone treatments, and the luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels are within the laboratory postmenopausal reference value range, also Can be considered post-menopausal;
  3. Have received irreversible sterilization, including hysterectomy, bilateral ovariectomy or bilateral fallopian tube resection, except for bilateral tubal ligation.
* For men, participants must agree to use appropriate methods of contraception or have been surgically sterilized during the trial period and 8 weeks after the last trial drug administration;

Exclusion Criteria:

* Patients who have previously received Anlotinib hydrochloride treatment or any anti-PD-1, anti-PD-L1, and anti-CTLA-4 antibody treatment;
* It is known that ESCC tends to be completely obstructed under endoscopy and requires interventional therapy to relieve the obstruction;
* ESCC patients with ulcer; Note: This mainly refers to patients whose ulcers are adjacent to blood vessels which increase the risk of bleeding.
* Patients who have received stent implantation in the esophagus or trachea;
* Patients who have a higher risk of bleeding or perforation due to the tumor's obvious invasion of the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed a fistula;
* Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before enrollment;
* There are a variety of factors that affect the use of therapeutic drugs, such as: inability to swallow or chronic diarrhea or intestinal obstruction, significantly affecting the administration and absorption of the drug, or a known history of severe allergies to any of the drug components in this study.
* The patient has received anti-tumor treatment with Chinese medicine in the past 2 weeks (Chinese medicine contains the following medicinal materials such as Brucea javanica, coix seed, lentinan, cantharidin, toad skin, astragalus, sophora flavescens, black bone vine, myrobalan, etc.), However, patients who took more than 2 weeks from the last anti-tumor treatment of Chinese medicine are allowed to join the group;
* The burden of liver metastases accounts for more than 50% of the entire liver volume;
* Patients with any severe and/uncontrolled diseases, including:

  1. Patients with poor blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg); or patients using two or more antihypertensive drugs to control blood pressure; previous hypertensive crisis or high Patients with blood pressure encephalopathy;
  2. Patients with grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc interval >450ms for men and >470ms for women) and congestive heart failure ≥2 (New York Heart Association (NYHA) classification), severe /Unstable angina) and patients who have undergone coronary/peripheral artery bypass surgery;
  3. Active or uncontrolled serious infection (≥CTCAE grade 2 infection), and those who are known to have active tuberculosis;
  4. Renal failure requires hemodialysis or peritoneal dialysis
  5. Liver diseases such as liver cirrhosis, decompensated liver disease, chronic active hepatitis;
  6. Poor control of diabetes (fasting blood glucose (FBG)>10mmol/L);
  7. Urine routine test shows that urine protein is ≥++, and the 24-hour urine protein quantification is confirmed to be >1.0 g;
* Long-term unhealed wounds or fractures;
* Patients with symptoms of hematemesis, hematochezia and daily bleeding ≥2.5mL, or any bleeding event ≥CTCAE level 3 within 3 months before screening, or any bleeding signs or medical history judged by the investigator to be unsuitable regardless of the severity Enrolled patients; or patients with abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), have bleeding tendency or are receiving thrombolytic or anticoagulant therapy; Note: Under the premise that the international normalized ratio of prothrombin time (INR) ≤ 1.5, the use of low-dose heparin (daily dosage for adults is 6,000 to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg);
* A history of gastrointestinal perforation and/or fistula in the 6 months before the enrollment treatment; or arterial/venous thrombotic events, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and lungs Embolizer
* Central nervous system metastases and/or cancerous meningitis with symptoms or active stages are known to exist;
* Ascites with clinical significance, including any ascites that can be found on physical examination, ascites that has been treated in the past or that still needs to be treated, and only those with a small amount of ascites but asymptomatic on imaging can be selected;
* Patients with moderate effusion in both pleural cavities, or large effusion in one pleural cavity, or patients who have caused respiratory dysfunction and need drainage;
* Suffer from interstitial lung disease that requires steroid therapy;
* Uncontrolled metabolic disorders or secondary reactions of other non-malignant tumor organs or systemic diseases or cancers, which may lead to higher medical risks and/or uncertainty in survival evaluation;
* Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders;
* Have a history of immunodeficiency, including those who have tested positive for HIV or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
* History of other primary malignant tumors, except for the following: a) Malignant tumors that have been completely remitted for at least 2 years before enrollment and no other treatment is required during the study period; b) Non-melanoma skin that has been adequately treated and has no evidence of disease recurrence Carcinoma or malignant freckle-like nevus; c) Carcinoma in situ that has been adequately treated and has no evidence of disease recurrence;
* Any of the following immune-related medical history and treatment history:

  1. There is any active autoimmune disease or a history of autoimmune disease (the following but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; subjects who require bronchodilators for medical intervention Asthma cannot be included); but the following patients are allowed to be included in the group: vitiligo, psoriasis, hair loss without systemic treatment, well-controlled type I diabetes, and hypothyroidism with normal thyroid function after replacement therapy;
  2. Diagnosed with immunodeficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose>10mg/day of prednisone or other curative hormones), and remain within 2 weeks before the first administration Continuing to use
  3. Have received any live vaccines, attenuated vaccines (including anti-infective vaccines, such as flu vaccines, varicella vaccines, etc.) or inactivated vaccines within 4 weeks before enrollment, and plan to vaccinate live vaccines/attenuated vaccines/inactivated vaccines during the study period Vaccine; used systemic immunostimulatory agents (including but not limited to interferon and IL-2) within 2 weeks before the start of the study treatment;
* During pregnancy or lactation, or planning to become pregnant during the study period or within 3 months after the last administration of TQB2450 or Anlotinib;
* According to the judgment of the investigator, there is a concomitant disease that seriously endangers the safety of the patient or affects the patient to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | about 2 years
  The RECIST1.1 and iRECIST standards were used to evaluate the efficacy of drugs, with the RECIST1.1 evaluation standard as the main and the iRECIST standard as a supplement.

SECONDARY OUTCOMES:
Safety:adverse events | about 2 years
  adverse events (AEs) categorized by severity in accordance with the NCI CTC AE Version 5.0
Progression Free Survival(PFS) | about 2 years
Disease Control Rate(DCR) | about 2 years
Duration of Response(DoR) | about 2 years
Overall Survival(OS) | about 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Anyang Tumour Hospital, Anyang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhumadian Central Hospital, Zhumadian

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meng X, Yang X, Hong Y, Wang W, Zhang Z, Xia J, Chen Y, Zhou Y, Lu T, Song M, Shan Z, Wu T, Wu W, Shen L, Guan L, Ma M, Wang L, Luo X, Xin D, Ma Y, Jiang G, Qi Y, Jiang B, Zhang D, Hu B, Wu X, Peng Z, Wang F. Anlotinib combined with benmelstobart as a chemo-free first-line treatment in advanced esophageal squamous cell carcinoma: an exploratory multicenter, single-arm phase II clinical trial. Mol Cancer. 2025 Jun 11;24(1):175. doi: 10.1186/s12943-025-02376-w. PMID 40500695